CLINICAL TRIAL: NCT00131261
Title: A Phase II Clinical Trial of PXD101 in Patients With Advanced Multiple Myeloma
Brief Title: Clinical Trial of PXD101 in Patients With Advanced Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PXD101-301-G
Record Dates: First submitted 2005-08-17; First posted 2005-08-18 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Neoplasms
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — belinostat; Dexamethasone

INTERVENTIONS:
Drug: PXD101
Drug: Dexamethasone

SUMMARY:
The purpose of this open-label, non-randomized trial is to assess the safety and effectiveness of PXD101, both alone and in combination with dexamethasone, in patients with advanced multiple myeloma. PXD101 is a new, potent histone deacetylase (HDAC) inhibitor. Various members of this class of drugs have shown activity in preclinical studies and in initial clinical trials of multiple myeloma and lymphoma. Furthermore, HDAC inhibitors, including PXD101, have been shown to sensitize myeloma cells to the killing effect of other chemotherapeutic agents, including dexamethasone, a well-established agent in relapsing myeloma.

ELIGIBILITY:
Inclusion criteria

1. Signed informed consent
2. A confirmed diagnosis of multiple myeloma, diagnostic criteria as follows, in patients who have failed at least two prior lines of therapy.

   Diagnostic criteria for multiple myeloma:

   A Monoclonal immunoglobulin (M-component) in serum of IgG-type > 30 g/l, of IgA type > 20 g/l, of IgD type or IgE type of any concentration and/or excretion of M-component in the urine of type k or l type > 1 g/24 hours.

   B M-component in serum and/or urine in lower concentration than indicated above in 'A'.

   C 10% or more plasma cells in bone marrow aspirate or plasmocytosis in biopsy from bone marrow or soft tissue tumor D Osteolytical bone lesions.

   The diagnosis of multiple myeloma demands one of the following combinations: A+C, A+D, or B+C+D.
3. Evaluable disease (as defined above)
4. Adequate bone marrow and hepatic functions including the following:

   1. WBC > 2.5 x 109/l, absolute neutrophil count ≥ 1.5 x 109/l, platelets ≥ 50x109/l
   2. Total bilirubin ≤1.5 x upper normal limit.
   3. AST (SGOT), ALT (SGPT) ≤2.5 x upper normal limit
5. Serum potassium within normal range.
6. Age ≥18 years
7. Performance status (PS) ≤2 (ECOG scale)
8. Estimated life expectancy greater than 3 months
9. Female patients with reproductive potential with a negative serum pregnancy test within the last 7 days before trial enrollment and use a safe contraceptive during and in a period of 60 days after the trial. Fertile female partners to male participants must likewise use contraceptive.

Exclusion criteria

1. Anticancer therapy including chemotherapy, radiotherapy, endocrine therapy, immunotherapy or use of other investigational agents within the last 4 weeks or a longer period depending on the defined characteristics of the agents used (e.g. 6 weeks for mitomycin or nitrosourea). Exception: bisphosphonates for bone disease caused by multiple myeloma.
2. Active infection or any medical condition likely to interfere with trial procedures.
3. Significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension, congestive heart failure related to primary cardiac disease, a condition requiring anti-arrhythmic therapy, ischemic or severe valvular heart disease, or a myocardial infarction within 6 months prior to the trial entry.
4. A marked baseline prolongation of QT/QTc interval, e.g., repeated demonstration of a QTc interval >500; Long QT Syndrome; the required use of concomitant medication on PXD101 infusion days that may cause Torsade de Pointes. (See Appendix B for list).
5. Patients with renal insufficiency defined as a calculated creatinine clearance of < 45 ml/min.
6. Clinically significant central nervous system disorders requiring neuroleptics or anti-convulsant medication.
7. Altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies
8. Other malignant diseases requiring treatment
9. Non-secretory multiple myeloma or symptomatic amyloidosis
10. Pregnant or breast-feeding women
11. Women of childbearing age and potential, who do not use effective contraception
12. Known HIV positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-01; Primary Completion 2007-01 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: enquiries@topotarget.com, Study Chair — Valerio Therapeutics
Locations (10):
- United States (4):
  - James Berenson, MD, Inc, West Hollywood, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Research Facility, New York, New York
- Rigshospitalet, Copenhagen, Denmark
- Norway (3):
  - Research Facility, Bergen
  - Research Facility, Oslo
  - Research Facility, Trondheim
- United Kingdom (2):
  - Christie Hospital NHS Trust, Manchester
  - The Royal Marsden NHS Trust, Surrey